CLINICAL TRIAL: NCT00682370
Title: Dose Escalation, Randomized, Placebo Controlled Study to Investigate the Effects of Intravenous Heme Arginate on Heme Oxygenase-1 (HO-1) and Heme Metabolism in Association With HO-1 Gene GTn Promoter Polymorphism in Healthy Male Subjects
Brief Title: Effects of Heme Arginate in Healthy Male Subjects
Acronym: HEMAHS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel Doberer (Other)
Responsible Party: Sponsor-Investigator, Daniel Doberer, Studienleiter, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT - 2007-003790-11
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Subjects; Heme Oxygenase; Genetic Polymorphism
MeSH Terms: interventions — Saline Solution; heme arginate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1 (Experimental): 0.3 mg/kg heme arginate
  Interventions: Drug: heme arginate
- A2 (Experimental): 1 mg/kg heme arginate
  Interventions: Drug: heme arginate
- A3 (Experimental): 3 mg/kg heme arginate
  Interventions: Drug: heme arginate
- P (Placebo Comparator): Placebo
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: saline solution — intravenous infusion, single dose
  Arms: P
Drug: heme arginate — intravenous infusion, single dose
  0.3 mg/kg heme arginate
  Arms: A1
Drug: heme arginate — intravenous infusion, single dose
  1 mg/kg heme arginate
  Arms: A2
Drug: heme arginate — intravenous infusion, single dose
  3 mg/kg heme arginate
  Arms: A3

SUMMARY:
Heme oxygenase 1 (HO-1) serves as a protective gene. It has been shown that one factor modulating HO-1 activity is a genetic variation in the HO-1 gene (functional GT length polymorphism in the promotor region). Heme arginate is a strong inducer of HO-1 as shown in several animal experimental studies. The aim of this clinical trial is to evaluate the HO-1 stimulation of heme arginate in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Male aged between 18 and 45 years (inclusive) at screening.
* No clinically significant findings on the physical examination at screening.
* Body mass index (BMI) between 18 and 28 kg/m2 (inclusive) at screening.
* 12-lead ECG without clinically relevant abnormalities at screening.
* Hematology, clinical chemistry, and urinalysis test results not deviating from the normal range to a clinically relevant extent at screening.
* Negative results from urine drug screen at screening.
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Known hypersensitivity to the study drug or any excipients of the drug formulation.
* Treatment with another investigational drug within 3 months prior to screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs.
* Smoking within the last 3 months prior to screening.
* Previous treatment with any prescribed or OTC medications (including herbal medicines such as St John's Wort) within 2 weeks prior to screening.
* Loss of 250 ml or more of blood within 3 months prior to screening.
* Positive results from the hepatitis serology, except for vaccinated subjects, at screening.
* Positive results from the HIV serology at screening.
* Presumed non-compliance.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The maximal HO-1 mRNA expression in PBMCs | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- See also: Department of Clinical Pharmacology, Medical University of Vienna — http://www.meduniwien.ac.at/klpharm/